CLINICAL TRIAL: NCT01000896
Title: A Phase I, Open-Label, Study to Assess the Safety, Tolerability, and Pharmacokinetics of Ascending Doses of AZD0530 in Combination With Carboplatin and Paclitaxel Chemotherapy in Japanese Patients With Advanced Solid Malignancies
Brief Title: Study to Assess Safety and Tolerability of AZD0530 in Combination With Carboplatin and Paclitaxel
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: AstraZeneca has discontinued the development of AZD0530. No new AstraZeneca-sponsored clinical studies will be initiated..
Sponsor: AstraZeneca (Industry)
Responsible Party: MSD, AstraZeneca
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D8180C00020
Record Dates: First submitted 2009-10-14; First posted 2009-10-23 (Estimated); Last update posted 2010-02-04 (Estimated); Status verified 2010-02

CONDITIONS: Cancer; Non Small Cell Lung Cancer; Epithelial Ovarian Cancer
Keywords: Phase I; cancer; solid tumors; advanced solid malignancies; NSCLC; epithelial ovarian cancer; dose escalation; combination treatment; src inhibitor; Japanese
MeSH Terms: conditions — Neoplasms; Carcinoma, Non-Small-Cell Lung; Carcinoma, Ovarian Epithelial | interventions — saracatinib; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AZD0530 + carboplatin and paclitaxel (Experimental): AZD0530 in combination with carboplatin and paclitaxel
  Interventions: Drug: AZD0530; Drug: Carboplatin; Drug: paclitaxel

INTERVENTIONS:
Drug: AZD0530 — film coated tablet, PO, daily
Drug: Carboplatin — intravenous, 3 weeks
  Other Names: Paraplatin
Drug: paclitaxel — intravenous, 3 weeks
  Other Names: Taxol

SUMMARY:
The primary purpose of this study is to explore the safety and tolerability of AZD0530 in combination with carboplatin and paclitaxel in Japanese patients with non small cell lung cancer and epithelial ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* Japanese patients with non small cell lung cancer or epithelial ovarian cancer
* Must be suitable for treatment with carboplatin and paclitaxel
* Relatively good overall health other than cancer

Exclusion Criteria:

* Poor bone marrow function (not producing enough blood cells).
* Poor liver or kidney function.
* Patients unable to discontinue drugs known to be potent inhibitors or inducers of CYP3A4 within 2 weeks prior to registration

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-09 (Estimated); Study Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
Assessment of adverse events (based on CTCAE version 3.0), laboratory values, vital sign measurements, general examination, HRCT, SpO2, ECG | Laboratory assessment prior to chemotherapy administration in all treatment cycles and on days 2, 8 and 15 in cycle 1. General exam, SpO2 and ECG prior to chemotherapy administration in all treatment cycles. HRCT scans performed days 21, 42, 70-98.

SECONDARY OUTCOMES:
Assessment of the pharmacokinetics of AZD0530 (Cssmax, Cssmin, tmax, AUCss0-24, CL/F), its N-desmethyl metabolite M594347 (Cssmax, Cssmin, tmax, AUCss0-24), and carboplatin / paclitaxel (Cmax, AUC, AUC0-t, t1/2, CL and Vss) | Schedule of PK assessment1. AZD0530/N-desmethyl metabolite M594347Cycle1-day21 -Cycle2-day2; 11point2. carboplatinCycle1-day1 ~ day2; 8 pointCycle2-day1 ~ day2; 8 point3. paclitaxelCycle1-day1 ~day2; 9 pointCycle2-day1 ~ day2; 9 point

CONTACTS AND LOCATIONS:
Overall Officials: Mary Stuart, Study Director — AstraZeneca; Takashi Seto, MD, PhD, Principal Investigator — National Hospital Organisation Kyushu Cancer Centre; Naoyuki Nogami, MD, Principal Investigator — National Hospital Organisation Shikoku Cancer Centre
Locations (2):
- Japan (2):
  - Research Site, Matsuyama, Ehime
  - Research Site, Fukuoka, Fukuoka